CLINICAL TRIAL: NCT05878600
Title: Targeted Cervical Spine Strengthening Exercises Versus Kendall Exercises in Patients With Forward Head Posture.
Brief Title: Cervical Spine Strengthening Exercises Versus Kendall Exercises in Patients With Forward Head Posture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0120
Record Dates: First submitted 2023-05-04; First posted 2023-05-26 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Forward Head Posture
Keywords: Forward head, Kendall exercises.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical spine strengthening group (Experimental): The participant will nod and chin tuck the head against the block with bands supporting the movement.
  An air-filled pressure cushion is placed under the occiput behind the cervical spine and conforms to the subject's shape. With a head nod, the pressure on the cuff increases and is shown by the dial. 10 repetitions of 5 seconds hold will be performed for 8 weeks and strength is measured by sphygmomanometer
  Interventions: Other: cervical spine strengthening
- Kendall exercise group (Active Comparator): patient is seated and the exercises are performed which include stretching pectoralis muscle, placing both hands on the occipital area and pulling the elbows back up and performing arm abduction and external rotation; and (2) strengthening shoulder retraction, Strengthening the deep cervical flexors and Stretching the cervical extensors
  Interventions: Other: kendall's exercise

INTERVENTIONS:
Other: kendall's exercise — comparative effect of targeted cervical spine strengthening versus kendalls exercise will be analyzed
  Other Names: cervical spine strengthening
  Arms: Kendall exercise group
Other: cervical spine strengthening — sole effect of cervical spine strengthening will be analyzed
  Arms: cervical spine strengthening group

SUMMARY:
To compare the effects of targeted cervical spine strengthening exercises and Kendall exercise in patients with forward head posture

DETAILED DESCRIPTION:
Studies have evaluated the effect of Kendall's exercises and found it effective for recovery. Studies have also concluded that targeted strengthening of flexors reverse the symptoms. The purpose of this study will elaborate either there is a difference in time taken to achieve normal head alignment between a targeted muscle that is prone to weakness or a technique that involves strengthening of weakened muscle plus stretching of shortened muscles. As there is a vast variety of correcting exercise program in the literature, the decision to choose the best option may be challenging. This study may help physiotherapists to apply treatment that is directly directing the main culprit.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 20-40 years with no signs of degeneration.
* Individuals having cranio-vertebral angle less than 50
* Those who have not gone under rehabilitation for last 6 months
* Those who are computer users for more than 3 hours a day or more.

Exclusion Criteria:

* Spinal trauma
* Musculoskeletal abnormality in the cervical spine
* Rheumatologic disorders
* Any bony or soft tissue systemic disease
* Congenital defects
* Disc pathology

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Change in NPRS | 8th week
  Pain intensity will be assessed by numeric pain rating scale NPRS. The 11-point NPRS (intervals from 0-10) is used to quantify pain intensity; 0 represents no pain, and 10 represent the worst possible agony. The NPRS is a valid and reliable instrument for older persons. Participants will be asked to select the number that most accurately describes their level of pain. At the baseline assessment, following each exercise session during the 8-week intervention, and finally at the end of the intervention Programmed, the NPRS scores will be recorded Changes from Basline to 8th week

SECONDARY OUTCOMES:
Range of motion | 8th week
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position. The long arm goniometers are more accurate for joints with long levers like the knee and hip joints. A universal goniometer has three parts. A body: It is designed like a protractor and may form a full or a half-circle. It has a scale for the measurement of the angle. The scale can extend either from 0 to 180 degrees or 180 to 0 degrees. A fulcrum: The screw-like device can be tightened to fix the moving arm in a particular position or loosened to permit free movement. The moving arm is the arm of the goniometer, which aligns with the mobile part of the joint measured.
  Changes from Basline to 8th week

OTHER OUTCOMES:
neck disability index | 8th week
  The neck disability index NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 50 Changes from Basline to 8th week
Photogrammetry | 8th week
  It is used for postural evaluation. Most common way to find forward head posture is y measuring craniovertebral angle. Photos were taken from patients' right side and analysis is done by using ImageJ software Changes from Basline to 8th week

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- The Bank of Punjab, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mylonas K, Angelopoulos P, Billis E, Tsepis E, Fousekis K. Combining targeted instrument-assisted soft tissue mobilization applications and neuromuscular exercises can correct forward head posture and improve the functionality of patients with mechanical neck pain: a randomized control study. BMC Musculoskelet Disord. 2021 Feb 21;22(1):212. doi: 10.1186/s12891-021-04080-4. PMID 33612123
- [Background] Handa Y, Okada K, Takasaki H. Lumbar Roll Usage While Sitting Reduces the Forward Head Posture in Healthy Individuals: A Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2021 May 13;18(10):5171. doi: 10.3390/ijerph18105171. PMID 34068139
- [Background] Baskurt Z, Baskurt F, Gelecek N, Ozkan MH. The effectiveness of scapular stabilization exercise in the patients with subacromial impingement syndrome. J Back Musculoskelet Rehabil. 2011;24(3):173-9. doi: 10.3233/BMR-2011-0291. PMID 21849731
- [Background] Shiravi S, Letafatkar A, Bertozzi L, Pillastrini P, Khaleghi Tazji M. Efficacy of Abdominal Control Feedback and Scapula Stabilization Exercises in Participants With Forward Head, Round Shoulder Postures and Neck Movement Impairment. Sports Health. 2019 May/Jun;11(3):272-279. doi: 10.1177/1941738119835223. Epub 2019 Apr 23. PMID 31013190
- [Background] Ravichandran H, Janakiraman B, Gelaw AY, Fisseha B, Sundaram S, Sharma HR. Effect of scapular stabilization exercise program in patients with subacromial impingement syndrome: a systematic review. J Exerc Rehabil. 2020 Jun 30;16(3):216-226. doi: 10.12965/jer.2040256.128. eCollection 2020 Jun. PMID 32724778
- [Background] Mahashabde R, Fernandez R, Sabnis S. Validity and reliability of the aneroid sphygmomanometer using a paediatric size cuff for craniocervical flexion test. Int J Evid Based Healthc. 2013 Dec;11(4):285-90. doi: 10.1111/1744-1609.12048. PMID 24298922
- [Background] Mahmoud NF, Hassan KA, Abdelmajeed SF, Moustafa IM, Silva AG. The Relationship Between Forward Head Posture and Neck Pain: a Systematic Review and Meta-Analysis. Curr Rev Musculoskelet Med. 2019 Dec;12(4):562-577. doi: 10.1007/s12178-019-09594-y. PMID 31773477
- [Background] Lee DY, Nam CW, Sung YB, Kim K, Lee HY. Changes in rounded shoulder posture and forward head posture according to exercise methods. J Phys Ther Sci. 2017 Oct;29(10):1824-1827. doi: 10.1589/jpts.29.1824. Epub 2017 Oct 21. PMID 29184298
- [Background] Fathollahnejad K, Letafatkar A, Hadadnezhad M. The effect of manual therapy and stabilizing exercises on forward head and rounded shoulder postures: a six-week intervention with a one-month follow-up study. BMC Musculoskelet Disord. 2019 Feb 18;20(1):86. doi: 10.1186/s12891-019-2438-y. PMID 30777064